CLINICAL TRIAL: NCT04988399
Title: Feasibility of Internet-based Reiki as an Intervention for Tinnitus
Brief Title: Internet-based Reiki for Tinnitus 2021
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn prior to Einstein IRB approval
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12737
Record Dates: First submitted 2021-07-16; First posted 2021-08-03 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Tinnitus
Keywords: Tinnitus; Reiki
MeSH Terms: conditions — Tinnitus | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reiki Recipients (Experimental): The Practitioner enters a gassho (two hands coming together at the heart) meditative state with the Distance Symbol. Reiji-ho - moving the joined hands until the thumbs touch the space between the brows. Going into a relaxed state by using a breathing technique. Say the person's name three times. Proceed with byosen (method using the sensitivity in the hands to treat those areas in need of Reiki) scanning technique. Chiryo (standard session visualizing all hand positions) for 5 minutes each: Jawbone-Back of the head-Throat-Lungs-Area of participant's concern-Stomach-Intestines-Kidneys-Spinal cord. At the end of the session, visualize towards the participant's feet to help integrate the healing. Visualize brushing the Biomagnetic field around the participant's body from head to feet. Inform the participant that the session has been completed. Include time to rest quietly for a few minutes. Encourage participant to sip water (if they prefer) and ask them about their experience.
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Reiki — Reiki is a wellness practice of energy healing that began in Japan and is now practiced throughout the world. The principle of Reiki is that everything in the universe consists of energy including the human body, and deviations of this energy can lead to disease (Doğan 2018). Reiki does not have a religious doctrine and is accepted by people of all backgrounds and belief systems (McManus, 2017, p. 1056). Reiki is considered by practitioners to be a great tool for stress reduction and relaxation (International Association of Reiki Practitioners). Many people use Reiki for wellness. Reiki is not a cure for a disease or illness, but it may assist the body in creating an environment to facilitate healing. According to the Center for Reiki Research, Reiki is an effective approach for reducing pain, depression, and anxiety. Tinnitus is a pain percept, and it is likely Reiki may reduce pain and anxiety in patients with tinnitus.

SUMMARY:
The objectives of the study will be 1) to develop and show the feasibility of an internet-based Reiki therapy as an intervention for tinnitus, 2) to deliver Reiki therapy for tinnitus as a potential treatment, 3) to maintain a meaningful cohort of participants over a 6-month protocol, and 4) to collect pilot data on the potential benefit of internet-based Reiki therapy on tinnitus-related quality of life. Patients will also be provided with information on other potential tinnitus therapies.

DETAILED DESCRIPTION:
Reiki is a wellness practice of energy healing that began in Japan and is now practiced throughout the world. The principle of Reiki is that everything in the universe consists of energy including the human body, and deviations of this energy can lead to disease. Reiki does not have a religious doctrine and is accepted by people of all backgrounds and belief systems. Reiki is considered by practitioners to be a great tool for stress reduction and relaxation (International Association of Reiki Practitioners).

Many people use Reiki for wellness. Reiki is not a cure for a disease or illness, but it may assist the body in creating an environment to facilitate healing. According to the Center for Reiki Research, Reiki is an effective approach for reducing pain, depression, and anxiety. Tinnitus is a pain percept, and it is likely Reiki may reduce pain and anxiety in patients with tinnitus.

The aims of the study are to show the feasibility of an internet-based Reiki therapy as an intervention for tinnitus. Home based therapy can reduce the stress of receiving therapy in an unfamiliar environment. Home-based therapy can also allow the participants to regain more control their surroundings, making them more likely to benefit from relaxation and stress relief benefits of Reiki.

Specific Aim 1: The first aim is to show that our Reiki therapy can be delivered to tinnitus patients on an internet-based platform This aim will be achieved if the investigators can recruit patients into the study and deliver internet-based therapy over the 6 months of the protocol while retaining a meaningful 30 percent of our cohort.

Specific Aim 2: The second aim is to show that participants perceive a benefit from the therapy protocol. This aim will be studied by retaining a meaningful cohort of participants and by analyzing data from the questionnaire results for the Tinnitus Handicap Inventory (THI) and Tinnitus Functional Index (TFI) before treatment, at 3 months and after 6 months of treatment and comparing them to the participants' baseline questionnaires. Data from the questionnaires will be used to determine sample size needed for a larger blinded control study.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking patients with unilateral or bilateral tinnitus

Exclusion Criteria:

* People under the age of 18
* People without internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Reported Tinnitus Relief | 6 months
  Change from baseline after Reiki treatment for tinnitus sufferers. Reduced stress in tinnitus sufferers seen as changes of the Tinnitus Handicap Inventory or Tinnitus Functional Index. Maximum possible score = 250 if the respondent were to rate all 25 TFI items at the maximum value of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Dinces, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No